CLINICAL TRIAL: NCT00279526
Title: Depression and Increased Health Services Utilization Among Elderly Primary Care Patients
Status: Completed | Type: Observational
Sponsor: Soroka University Medical Center (Other)
Other Study IDs: sor417105ctil
Record Dates: First submitted 2006-01-18; First posted 2006-01-19 (Estimated); Last update posted 2007-05-25 (Estimated); Status verified 2007-05

CONDITIONS: Depression
Keywords: Depression; Health services utilization; Elderly; Primary Care
MeSH Terms: conditions — Depression; Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Other

SUMMARY:
The increase in life expectancy in the 21st century has resulted in a major growth in the prevalence of age-related diseases and conditions. Depression has been found to be the most prevalent among the various mental disorders in later life. It was emphasized that depression in the elderly is a persistent or recurrent disorder resulting from psychosocial stress or physiologic effects of disease and can lead to disability, cognitive impairments, intensified symptoms of other medical conditions and increased utilization of health care services. Due to the rapidly aging population, depression is a serious public health concern that has a great impact on quality of life and may lay a considerable burden on the health care systems. However depression among the elderly may prove to be hard to diagnose since in aged persons depressive symptoms are often masked by somatic complaints or by cognitive impairments. Consequently depression is often under diagnosed and the patients continue to visit constantly the nurse or the physician without getting an adequate answer to their problem. For that reason over utilization of health care services may be an indicator to the presence of undiagnosed depression. The purpose of this study is to examine the relationships between socio-demographic variables, high primary care utilization and depressive symptomatology among aged patients.

DETAILED DESCRIPTION:
Introduction The number of Israel's elderly (65 plus) has increased from just 85,200 (4.8% of the population) in 1955 to approximately 670,000 people (about 10%) in 2003 (Brodsky et al., 2005). According to the most conservative of three projections offered by the Israeli Central Bureau of Statistics (CBS), the number of seniors is expected to be approximately 676,500 (9.8% of the population) in 2005, to rise to 722,500 people (10.7% of the population) by 2010 and increase to 1,025,800 (almost 12% of the population) by the year 2020.

The increase in life expectancy in the 20th century has resulted in a major growth in the prevalence of age-related diseases and conditions. Depression has been found to be the most prevalent among various mental disorders in later life and is the third most common reason for consultation in primary care (Shah, 1992). Research shows that 10-15% of the persons over 65 years of age suffer from various levels of depressive symptoms (Jacob& Palmer, 1998).

Sadock & Sadock (2003) state that depression among elderly may reach up to 15 percent and among these suffering from dementia from 25- 50 percent. Israeli studies show similar rates of depressive symptomatology as performed in other Western countries. A prevalence of 21.5 percent of depressive symptomatology was found among a random sample of 937 Israeli adults. (Iancu et al., 2003).

Depression represents a heterogeneous set of disorders, usually characterized by sad mood and inability to experience pleasure. Among the elderly it often may present itself atypically, with somatic symptoms dominating the clinical picture (Jacob & Palmer, 1998). Common physical complaints, start with the most common features as loss of energy or fatigue, unexplained pain, gastrointestinal symptoms, headache, dizziness, palpitations, heartburn, numbness, loss of appetite, insomnia specifically early morning awakening. In general, the more unexplained somatic complaints and physical symptoms a patient have, the higher the likelihood of depression (Glass 2003). Elderly depression impairs significantly the quality of life by leading to disability, cognitive impairments, intensified symptoms from medical conditions and increases utilization of health care services and the direct and indirect medical costs (Luber et al., 2001).

Herrman et al.,( 2002) argue that health care utilization among depressed patients is higher then among those without depression. Elderly with depressive symptoms found to be at least as twice as likely to use emergency department and medical inpatient hospital services compared to patients without depressive symptomatology ( Himelhoch et al., 2002). Simon & Ormel(1995) as well as Katon et al. (2003) stated that patients with depressive symptoms account for 43-52% higher health care costs than patients without depressive symptoms.

The increase in costs associated with depressive symptoms was noted even after adjusting for the severity of chronic medical illness (Glass, 2003). According to the WHO the significance of illness burden attributable to depression increases with age and thus will grow further by the year 2020 based upon projected demographic shifts towards an older population (Peveler et al., 2002).

This trend was showed in Israel by Brodsky et al.( 2005). They reported an elderly average of 11.5 visits at the FP per year while, in the USA, only 25% of the elderly population visited any physician 10 or more times annually - including visits to the ER and home visits (Health, United States,2003).

Consequently detecting and treating elderly patients with depressive symptoms in Israel, may be cost-effective and produce improvement in health and well-being for the money spent in the care of these older adults.

However depression in the aged patient may be atypical in nature and more difficult to diagnose from that in the general population. Therefore it is often under-diagnosed and under-treated (Jacob & Palmer, 1998). In contrast to younger depressed patients, elderly patients often avoid reporting or showing that their mood level and tend to hide their state of disease or, worse, they lack the consciousness of the disease and think that enjoying life less than before is an inevitable consequence of aging. Moreover, elderly sometimes attribute their depressive symptoms to general medical conditions. Other factors that may hinder distinguishing depression from other conditions are also concomitant diseases, especially dementia, polypharmacy and drug reactions (Glass, 2003). Furthermore Hybels et al. (2001) compared in their study the demographic and risk factor profiles of elderly individuals with less and more severe depression. The obtained results indicated the need to recognize that elderly adults who do not meet the Diagnostic and Statistical Manual of Mental Disorders (DSM) criteria for depression, and those who fall below the threshold on instruments such as the Center for Epidemiologic Studies-Depression scale (CES-D), may still experience depressive symptomatology that warrant attention.

The current scales used today measure physical deterioration as part of the depressive state, while among the older people these are part of the aging process and may confuse the therapist. The Geriatric Depression Scale (GDS) is a more specific tool for the measurement in this age group. It was developed during the 80's (Brink et al., 1982) proven valid and reliable at 1986 and was translated to many languages including Hebrew. (Zalsman et al., 1998). Today it is one of the most widely used instruments for the screening of depression among the elderly population.

To simplify the screening process a Yale Task Force on Geriatric Assessment has recommended the use of a single question, "Do you often feel sad or depressed?" (Lachs et al., 1990). Mahoney et al.( 1994 ) found this question as a valid and reliable short-form alternative.

In conclusion depression is a prevalent mental disorder in later life and a considerable impending public health problem since it may lay unnecessary cost burden on one hand and is difficult to diagnose on the other. Consequently, there is a need to find the most effective ways for early detection of this condition. This study will examine the question whether high health care services utilization and/ or sociodemographic background may predict the presence of depression among aged patients.

Objectives:

The purposes of this study is to examine the relationships between socio-demographic variables, comorbidity, depressive symptomatology and high primary care utilization.

METHOD:

Participants:

The study will be conducted in 10 primary health care clinics in urban communities of Beersheva, Israel. According to the average health care utilization, 11.5 visits to the FP per year (Brodsky et al., 2005)) among elderly in Israel, we classify two groups: "low care utilizers" with ≤ 6 visits per year and "high care utilizers" with ≥ 16 visits. Primary lists of "high and low care utilizer" will be obtained by query to "Clicks" electronic medical chart system ( Roshtov Soft wear industry ltd.) .

ELIGIBILITY:
Inclusion Criteria:-

* Age 65 or older,
* Clalit health organization client
* Outpatient
* Hebrew or English or Russian speaker
* Living in Beer Sheva

Exclusion Criteria:

* Known diagnosis of depression, major depression, bipolar disorder, psychosis, dementia or substance abuse
* Current acute illness

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 450
Dates: Start 2006-04; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yan Press, MD, Principal Investigator — Ben-Gurion University of the Negev
Locations (1):
- Department of Family Medicine, Faculty of Health Sciences, Ben Gurion University of the Negev, Beersheba, Israel